CLINICAL TRIAL: NCT00408577
Title: Prevention of Cardiovascular Relapses by L-Arginine Oral Administration in Patients With CAD and IGT and/or Insulin Resistance.
Brief Title: Prevention of Cardiac and Vascular Events in Patients With NGT/IGT.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OSRAFFA_III_2004_003
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Cardiovascular Disease
Keywords: glucose intolerance; cardiovascular disease; insulin resistance; endothelial dysfunction
MeSH Terms: conditions — Cardiovascular Diseases; Glucose Intolerance; Insulin Resistance | interventions — Arginine

INTERVENTIONS:
Drug: L-arginine

SUMMARY:
Impaired glucose tolerance or mild glucose elevations in the non-diabetic range are associated with increased cardiovascular disease and recent studies suggested the need to detect these glucose abnormalities early in the post-infarction period. Although in the last ten years procedures of coronary revascularisation have dramatically improved the outcome of non diabetic patients affected by ischemic heart disease, these procedures are less effective in patients with type 2 diabetes mellitus and IGT. Possible causes of worse prognosis in these patients could be related to the presence of hyperinsulinemia and insulin resistance due to the well known effect of insulin to increase neointimal tissue proliferation and in-stent restenosis, by stimulating vascular smooth muscle cell growth factors and migration. In addition, it is well known that endothelial dysfunction is an early functional disturbance in the development of atherosclerotic lesions. The impairment of eNOS action might change the turnover rate of eNOS or nitric oxide production and action influencing nitric oxide signalling, apoptosis cascade and angiogenesis. All these factors can contribute to endothelial dysfunction to a certain extent, and accelerate atherosclerosis with increased risk for cardiovascular disease.

The constitutively expressed eNOS, is likely to be the major contributors to whole-body nitric oxide production. It is interesting to note that a region of chromosome 7q seems to influence both insulin resistance and blood pressure, suggesting that this locus may broadly influence traits associated with insulin resistance.

L-arginine is an essential amino acid and its availability is important for the normal endothelial cell function and its intracellular reduction may contribute to the dysfunctional endothelial state. It is well known that L-arginine is as a precursor for nitric oxide and both in vitro and in vivo studies have demonstrated that L-arginine can augment vascular dilation under certain conditions.

Our hypothesis is to evaluate the modulating effect of L-arginine on metabolic, endothelial variables and on myocardial function in patients with cardiovascular disease.

DETAILED DESCRIPTION:
Condition: Patients submitted to coronary revascularization characterized for glucose tolerance after OGTT Intervention: L-arginine for 6 months Inclusion criteria: patients in stable clinical conditions after coronary revascularization (CABG and percutaneous angioplasty with/without stent implantation). Age > 30 years, male and female. Fasting glucose levels below 126 mg/dl.

Exclusion criteria. Type 1 diabetes mellitus, known type 2 diabetes mellitus, pregnancy, impaired kidney and liver function, severe and not treated arterial hypertension.

Study type: randomized, double blind, Placebo, parallel

ELIGIBILITY:
Inclusion Criteria:

* patients in stable clinical conditions after coronary revascularization (CABG and percutaneous angioplasty with/without stent implantation).
* Age > 30 years, male and female.
* Fasting glucose levels below 126 mg/dl.

Exclusion Criteria:

* Type 1 diabetes mellitus,
* known type 2 diabetes mellitus,
* pregnancy,
* impaired kidney and liver function,
* severe and not treated arterial hypertension.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-11; Study Completion 2006-11

PRIMARY OUTCOMES:
Evaluation of 6 months L-arginine/placebo oral treatment on glucose tolerance and insulin resistance measured by OGTT

SECONDARY OUTCOMES:
Evaluation of 6 months L-arginine/placebo oral treatment on endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: PierMarco Piatti, MD, Principal Investigator — Scientific Institute San Raffaele
Locations (1):
- Scientific Institute San Raffaele, Milan, Milan, Italy